CLINICAL TRIAL: NCT05512286
Title: Comparison of Patient-Reported Outcome and Safety Outcomes Between Preoperative and Postmastectomy Radiotherapy in Breast Cancer Patients with Reconstruction of DIEP Flap: a Multicenter，Prospective，Open-label，Randomized Controlled Trial
Brief Title: Patient-Reported Outcome and Safety Between Preoperative and Postmastectomy Radiotherapy in DIEP Flap Reconstruction
Acronym: CAPPELLA
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Fudan University (Other)
Collaborators: Huashan Hospital (Other); Hunan Cancer Hospital (Other); Cancer Hospital of Guangxi Medical University (Other); Yunnan Cancer Hospital (Other); Zhejiang Cancer Hospital (Other); Henan Cancer Hospital (Other Government)
Responsible Party: Principal Investigator, Jiong Wu, Professor, Fudan University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CBCSG041
Record Dates: First submitted 2022-08-19; First posted 2022-08-23 (Actual); Last update posted 2024-11-25 (Actual); Status verified 2024-11

CONDITIONS: Breast Cancer
Keywords: DIEP flap; radiotherapy; breast cancer
MeSH Terms: conditions — Breast Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Preoperative radiotherapy (Experimental): Radiotherapy followed by mastectomy and DIEP flap reconstruction
  Interventions: Radiation: Preoperative radiotherapy
- Postmastectomy radiotherapy (Active Comparator): Radiotherapy after mastectomy and DIEP flap reconstruction
  Interventions: Radiation: Postmastectomy radiotherapy

INTERVENTIONS:
Radiation: Preoperative radiotherapy — Radiotherapy followed by mastectomy and DIEP flap reconstruction
  Arms: Preoperative radiotherapy
Radiation: Postmastectomy radiotherapy — Radiotherapy after mastectomy and DIEP flap reconstruction
  Arms: Postmastectomy radiotherapy

SUMMARY:
This study is the first prospective randomized study assessing the patient-reported outcomes and safety outcomes between preoperative and postmastectomy radiotherapy in locally advanced breast cancer patients with immediate reconstruction of deep inferior epigastric perforator(DIEP) flap. Radiotherapy before mastectomy and autologous free-flap breast reconstruction can avoid adverse radiation effects on healthy donor tissues and delays to adjuvant radiotherapy. We aimed to explore the feasibility of preoperative radiotherapy followed by DIEP flap reconstruction in patients with breast cancer requiring mastectomy.

ELIGIBILITY:
Inclusion Criteria:

* Patients with histological proven invasive breast cancer;
* Clinical T0-3, T4b and N0-3a disease who require neoadjuvant chemotherapy;
* No distant metastasis;
* Adjuvant radiotherapy and who are suitable for DIEP flap reconstruction at the time of mastectomy.

Exclusion Criteria:

* Patients enrolled in other clinical trial which may as influence the outcome;
* Patients received neoadjuvant therapy without radiotherapy indications；
* Disease progression during neoadjuvant chemotherapy；
* Patients of pregnancy or lactation；
* Previous history of diabetes；
* Previous history of heavy smoking.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Estimated)
Dates: Start 2022-08-25 (Actual); Primary Completion 2026-07-01 (Estimated); Study Completion 2027-10-01 (Estimated)

PRIMARY OUTCOMES:
Patient satisfaction with breasts questionnaire Patient satisfaction of breast | 24 months after surgery
  Patient satisfaction with breasts (as measured using the BREAST-Q reconstruction module) 24 months after surgery.

SECONDARY OUTCOMES:
Complications of surgery | 3 months, 12 months, and 24 months
  Complications of surgery
Complications of radiotherapy | 3 months, 12 months, and 24 months after radiotherapy
  Complications of radiotherapy
Failure rate of breast reconstruction surgery | 8 weeks after surgery
  Failure rate of breast reconstruction surgery
Patient satisfaction with outcome questionnaire | 3months, 12 months, and 24 months after surgery
  Patient satisfaction with outcome (as measured using the BREAST-Q reconstruction module) 3months, 12 months, and 24 months after surgery
Aesthetic evaluation | 12 months and 24 months after surgery
  Aesthetic evaluation (as measured using the Harris Score) 12 months and 24months after surgery. Breast aesthetic evaluation will subjectively be evaluated by two experts who applied the Harris score giving a mark of 1-4 for a poor to excellent result.
Total pathologic complete response (tpCR) | up to 4 weeks after surgery
  pathologic complete response of breast and lymph nodes
3-year disease free survival (DFS) | 3 years after diagnosis
  Oncological safety

CONTACTS AND LOCATIONS:
Overall Officials: Jiong Wu, Principal Investigator — Fudan University
Locations (6):
- China (6):
  - Guangxi Provincial Cancer Hospital, Nanning, Guangxi
  - Henan Provincial Cancer Hospital, Zhengzhou, Henan
  - Hunan Provincial Cancer Hospital, Changsha, Hunan
  - Huashan Hospital of Fudan University, Shanghai, Shanghai Municipality
  - Yunnan Provincial Cancer Hospital, Kunming, Yunnan
  - Zhejiang Provincial Cancer Hospital, Hangzhou, Zhejiang

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Hao S, Hou J, Zhang L, Zhou C, Hou Y, Yu K, Hu Z, Liu G, Di G, Shao ZM, Yu X, Wu J. Protocol for a multicentre, prospective, open-label, randomised controlled trial to compare PROs and safety outcomes between preoperative and postmastectomy radiotherapy in locally advanced breast cancer patients with immediate reconstruction via a deep inferior epigastric perforator flap (CAPPELLA) in China. BMJ Open. 2025 Jan 20;15(1):e086980. doi: 10.1136/bmjopen-2024-086980. PMID 39832996